CLINICAL TRIAL: NCT06342245
Title: Low-temperature Radiofrequency Coblation Micro-tenotomy for the Treatment of Achilles Tendinopathy; a Multicentre, Prospective, Randomized Controlled Clinical Trial.
Brief Title: Low-temperature Radiofrequency Coblation Micro-tenotomy for the Treatment of Achilles Tendinopathy
Acronym: AT RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.568
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Intervention Model Description: This is a multicentre prospective randomized, double-blinded, placebo-controlled superiority trial with two parallel groups and a 1:1 allocation ratio to investigate the effectiveness of radiofrequency coblation micro-tenotomy for patients with Achilles tendinopathy. All participants will be randomized into two groups: the intervention group (n=24; radiofrequency coblation micro-tenotomy + endoscopic Achilles debridement) and the control group (n=24; endoscopic Achilles debridement only).
  Investigators will obtain written consent from all participants before the commencement of this study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency coblation micro-tenotomy + endoscopic Achilles debridement (Experimental): The patient will lie prone on the surgical table, and the area of tendinopathy will be visualized with endoscopy. Endoscopic-assisted creation of a percutaneous mesh (quincunx) pattern of 1mm skin incisions will be made over the area of tendinopathy with a 5mm distance between each incision. Radiofrequency micro-tenotomy with low-temperature controlled ablation will be performed with the TOPAZ (Smith and Nephew) wand, which has a 1mm tip, and full thickness 1mm RF tendon debridement at 5mm intervals will be performed. Incisions will be fixed with sterile strips
  Interventions: Radiation: Radiofrequency coblation micro-tenotomy
- endoscopic Achilles debridement only (No Intervention): Minimally invasive and endoscopic procedures yield lower complication rates with similar patient satisfaction compared to open procedures. Minimally invasive and endoscopic procedures were recommended as the future surgical treatment of Achilles midportion tendinopathy.
  Both the control and the intervention group will undergo endoscopic Achilles tendon debridement. The procedure will be performed in the operating theatre under general or regional anesthesia. The patient will lie prone on the operating table, and the leg will be prepared and draped under sterile technique. Two co-axial 0.5cm endoscopic portals will be created as per standard protocol, and a 4mm scope will be introduced for visualization.

INTERVENTIONS:
Radiation: Radiofrequency coblation micro-tenotomy — Radiofrequency micro-tenotomy with low-temperature controlled ablation will be performed with the TOPAZ (Smith and Nephew) wand, which has a 1mm tip, and full thickness 1mm RF tendon debridement at 5mm intervals will be performed.
  Arms: radiofrequency coblation micro-tenotomy + endoscopic Achilles debridement

SUMMARY:
This is a prospective randomized, double-blinded, placebo-controlled superiority trial with two parallel groups and a 1:1 allocation ratio to investigate the effectiveness of radiofrequency coblation micro-tenotomy for patients with Achilles tendinopathy. All participants will be randomized into two groups: the intervention group (n=24; radiofrequency coblation micro-tenotomy + endoscopic Achilles debridement) and the control group (n=24; endoscopic Achilles debridement only). Adults (age >18) with clinically diagnosed midportion Achilles tendinopathy will be recruited and scheduled for ultrasound screening. All participants will undergo a 12-week eccentric exercise program taught by a registered physiotherapist / athletic trainer. Undergo Endoscopic Achilles debridement and Radiofrequency coblation micro-tenotomy intervention. Criteria for discontinuing or modifying allocated interventions, Strategies to improve adherence to interventions, Relevant concomitant care permitted or prohibited during the trial and Provisions for post-trial care. Outocme measure will use VISA-A, pain scores, ultrasound measurement of thickness and vascularity, calf muscle strength, and ankle range of motion.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion is ultrasound-confirmed Achilles tendinopathy. Adults (age >18) with clinically diagnosed midportion Achilles tendinopathy will be recruited and scheduled for ultrasound screening. Ultrasonography diagnostic criteria include a thickened Achilles tendon and a Colour Doppler of at least 1 out of 3 in the Öhberg score 2-6 cm proximal to the Achilles tendon insertion. Victorian Institute of Sports Assessment -Achilles (VISA-A) scores below 60 points.

Exclusion Criteria:

* Patients will be excluded if they had a history of major injury or surgery on the affected lower limb in the past year and have mental/physical limitations hindering the participant's ability to complete assessments (ankle arthritis, neuromuscular disorders, etc.), including severe cognitive impairment and psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-11 (Estimated); Primary Completion 2027-06-10 (Estimated); Study Completion 2027-06-11 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment | 2weeks, 4 weeks, 2 months, 3 months, 6 months, 1 yesr after sugery
  The primary outcome measure will be the Victorian Institute of Sports Assessment - Achilles (VISA-A) questionnaire, either the original English version or the validated Chinese version, depending on the participant's native tongue.

IPD SHARING:
Plan to Share IPD: No